CLINICAL TRIAL: NCT00954044
Title: Exercising Together: An Intervention for Prostate Cancer Survivors and Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5366
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: randomized clinical trial; prostate cancer; partnered exercise
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercising Together (Experimental): Partnered progressive resistance exercise
  Interventions: Behavioral: Randomized Exercise Intervention
- Usual Care (Placebo Comparator): Usual Care Control
  Interventions: Behavioral: Randomized Exercise Intervention

INTERVENTIONS:
Behavioral: Randomized Exercise Intervention — The Exercising Together training group will participate in 6 months of supervised, progressive partnered resistance exercise.
  Couples will participate in 2 exercise sessions a week for 6 months.
  Arms: Exercising Together
Behavioral: Randomized Exercise Intervention — Couples will continue doing their usual daily activities for 6 months
  Arms: Usual Care

SUMMARY:
The purpose of this study is to explore the benefits of "Exercising Together"-a partnered strength training program for married couples coping with prostate cancer- on the physical and emotional health of prostate cancer survivors and their spouse and on marital quality.

ELIGIBILITY:
Inclusion Criteria For PCS:

* Received treatment for histologically confirmed prostate cancer
* Not currently undergoing radiation therapy or chemotherapy for prostate cancer
* Currently residing with an identifiable spouse willing to participate
* 60 years and older at enrollment

Inclusion Criteria for Spouses:

* Currently residing with prostate cancer survivor

Exclusion Criteria for prostate cancer survivor and Spouses:

* Current participation in moderate/vigorous intensity resistance training 2 or more hours per week
* Cognitive difficulties that preclude answering the survey questions, participating in performance tests, or giving informed consent
* Medical condition, movement or neurological disorder, or medication that contraindicates participation in resistance exercise
* Unwillingness to be randomized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Physical function | baseline, 3, 6 months

SECONDARY OUTCOMES:
Marital quality | 0,3,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, PhD, Principal Investigator — Oregon Health & Science University-School of Nursing; Jessica Dobek, MS, Study Director — Oregon Health & Science University-School of Nursing
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Winters-Stone KM, Lyons KS, Bennett JA, Beer TM. Patterns and predictors of symptom incongruence in older couples coping with prostate cancer. Support Care Cancer. 2014 May;22(5):1341-8. doi: 10.1007/s00520-013-2092-0. Epub 2013 Dec 17. PMID 24337765
- [Derived] Winters-Stone KM, Lyons KS, Dobek J, Dieckmann NF, Bennett JA, Nail L, Beer TM. Benefits of partnered strength training for prostate cancer survivors and spouses: results from a randomized controlled trial of the Exercising Together project. J Cancer Surviv. 2016 Aug;10(4):633-44. doi: 10.1007/s11764-015-0509-0. Epub 2015 Dec 29. PMID 26715587